CLINICAL TRIAL: NCT03096496
Title: Long-term Quality of Life Symptom Burden in Acute Promyelocytic Leukemia (APL) Patients Treated With Arsenic Trioxide (ATO) or Standard Chemotherapy
Brief Title: Long-term QoL in Acute Promyelocytic Leukemia Treated With ATO or Standard Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: QoL-APL0816
Record Dates: First submitted 2017-01-24; First posted 2017-03-30 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Quality of life; acute promyelocytic leukemia; ATO
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GIMEMA APL0406 patients: APL survivors previously enrolled in GIMEMA APL0406 clinical trial and in 1st molecular CR after third consolidation treatment.
  Interventions: Other: QoL questionnaires

INTERVENTIONS:
Other: QoL questionnaires — Quality of life questionnaires

SUMMARY:
This is a prospective and international observational study run by the GIMEMA. All data will be centrally collected and analyzed at the GIMEMA Data Center in Rome (Italy). Patients reported outcomes will be collected using internationally validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* APL survivors enrolled in GIMEMA APL0406 clinical trial and in first molecular CR after third consolidation treatment
* Written informed consent.

Exclusion Criteria:

* APL patients previously enrolled in GIMEMA APL0406 trial who cannot be reached or who are lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously enrolled in a phase III randomized controlled trial that compared the efficacy and toxicity of standard ATRA plus chemotherapy versus ATRA plus ATO in low-intermediate risk APL patients.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
To examine cross-sectional long-term differences in health outcomes after treatment end. | Two years after study entry.
  Indicated by selected key-QoL outcomes (i.e. Fatigue, Cognitive and Role functioning scales from the EORTC-QLQ-C30 questionnaire), between APL patients treated with ATRA plus chemotherapy versus patients treated with ATRA plus ATO.

SECONDARY OUTCOMES:
To examine long-term differences in health outcomes after treatment end indicated by all QoL outcomes not considered in primary objectives, between APL patients treated with ATRA plus chemotherapy versus patients treated with ATRA plus ATO. | Two years after study entry.
  (including the functional status and symptomatology).
To investigate clinical, laboratory, socio-demographic and QoL factors predicting long-term health/QoL outcomes of APL patients after treatment end. | Two years after study entry.
  (as reported at 3rd consolidation).
To compare the long-term QoL profile, after treatment end, of APL patients treated with ATRA- chemotherapy and ATRA-ATO with that of their peers in the general population. | Two years after study entry.
  Compared with the general population (without cancer).
To assess and compare the cumulative incidence and types of physician-reported late adverse effects (e.g. cardiac function) and secondary cancer, between randomized treatment groups. | Two years after study entry.
  (ATRA plus chemotherapy versus ATRA plus ATO).
To assess and compare the prevalence of long-term patient-reported comorbidities and symptoms, after treatment end, between randomized treatment groups. | Two years after study entry.
  (ATRA plus chemotherapy versus ATRA plus ATO).

OTHER OUTCOMES:
To assess long-term QoL patterns over time of long-term APL survivors. | Two years after study entry.
  After treatment end, overall and by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Efficace, Study Chair — GIMEMA Foundation
Locations (16):
- Italy (16):
  - UOC Ematologia e Terapia Cellulare - Ospedale C. e G. Mazzoni di Ascoli Piceno, Ascoli Piceno
  - Spedali Civili - Brescia - Azienda Ospedaliera - U.O. Ematologia, Brescia
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze MEdiche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Cona
  - AOU - Policlinico G. Martino Messina Medicine Specialistiche e Oncologia Medica - UOC Ematologia, Messina
  - Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia - Padiglione Marcora 2do piano, Milan
  - UO Ematologia e Trapiano di Midollo - Ist. Scientifico Ospedale San Raffaele, Milan
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - SCDU Medicina Interna a indirizzo ematologico, Orbassano
  - U.O. di Oncoematologia -plesso ospedaliero "A. Tortora" di Pagani, Pagani
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ematologia - Dipartimento di Medicina Clinica e Sperimentale, Sassari
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino

REFERENCES:
- [Derived] Efficace F, Sparano F, Breccia M, Greco C, Carluccio P, Borlenghi E, Salutari P, Levato L, Baldi T, Mancini V, Finizio O, Autore F, Fazi P, Platzbecker U, Vignetti M, Voso MT. Health-related quality of life benefits of arsenic trioxide in patients with non-high-risk acute promyelocytic leukemia are sustained over time: long-term results of the GIMEMA APL0406 trial. Ann Hematol. 2024 Dec;103(12):5341-5349. doi: 10.1007/s00277-024-06038-7. Epub 2024 Oct 23. PMID 39438322
- [Derived] Efficace F, Platzbecker U, Breccia M, Cottone F, Carluccio P, Salutari P, Di Bona E, Borlenghi E, Autore F, Levato L, Finizio O, Mancini V, D'Ardia S, Schlenk RF, Melillo L, Fumagalli M, Fiedler W, Beltrami G, Fracchiolla NS, Bernardi M, Fazi P, Annibali O, Mayer K, Voso MT, Vignetti M. Long-term quality of life of patients with acute promyelocytic leukemia treated with arsenic trioxide vs chemotherapy. Blood Adv. 2021 Nov 9;5(21):4370-4379. doi: 10.1182/bloodadvances.2021004649. PMID 34529768
- See also: GIMEMA Foundation website — http://www.gimema.it